CLINICAL TRIAL: NCT00736073
Title: A Randomized, Double-Blind, Prospective Trial of Oral Administration of Aprepitant For Prevention of Post-Endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis
Brief Title: A Trial of Aprepitant For Prevention of Post-Endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00005149
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatitis
Keywords: pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): aprepitant
  Interventions: Drug: aprepitant
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: aprepitant — one dose of aprepitant (125 mg PO 4 hours) prior to their ERCP and one dose (80 mg PO) 18 hours after the first dose
  Arms: 1
Drug: Placebo — one dose of placebo (125 mg PO 4 hours) prior to their ERCP and one dose (80 mg PO) 18 hours after the first dose
  Arms: 2

SUMMARY:
The purpose of this study is to determine if giving Aprepitant 4 hours before and for two days after ERCP decreases the risk of developing pancreatitis after ERCP.

DETAILED DESCRIPTION:
This study involves taking a drug Aprepitant by mouth 4 hours before the ERCP and once a day for two days after the ERCP, in an attempt to reduce the risk of pancreatitis caused by ERCP. Pancreatitis, or injury and inflammation of the pancreas, is the most common complication of ERCP and occurs in approximately 6 out of every 100 patients undergoing ERCP. It may result in pain and lead to hospitalization and, in some cases, a need for further procedures such as surgery.

Aprepitant is a medication that is currently used to prevent nausea and vomiting in some patients caused by chemotherapy for the treatment of cancer. It is also approved for the prevention of post-operative nausea and vomiting. There is theoretical evidence from animal studies that the way in which Aprepitant works in the body may prevent pancreatitis.

ELIGIBILITY:
Inclusion Criteria: Patients selected for the study will be those undergoing ERCP who are at high risk for development of post-ERCP pancreatitis

* patients expected to undergo a sphincterotomy
* patients with suspected sphincter of oddi dysfunction
* patients with a known history in the past of post-ERCP pancreatitis
* patients less than 60 years of age

Exclusion Criteria:

* active pancreatitis
* if they are pregnant
* known adverse reaction to aprepitant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Poleski, MD, Principal Investigator — Duke University Medical Center, Department of Medicine, Division of Gastroenterology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects scheduled for ERCP as outpatient procedure in Duke clinic between Aug 2007 and October 2009
Pre-assignment Details: Investigational product to be given 4 hours before procedure
Groups:
- Arm 1-medication Pre and Post Procedure: Aprepitant
  aprepitant : one dose of aprepitant (125 mg PO 4 hours) prior to their ERCP and one dose (80 mg PO) 18 hours after the first dose
- Arm 2-Randomized to Placebo: Placebo
  Placebo : one dose of placebo (125 mg PO 4 hours) prior to their ERCP and one dose (80 mg PO) 18 hours after the first dose
Period: Overall Study
Arm/Group | Arm 1-medication Pre and Post Procedure | Arm 2-Randomized to Placebo
Started | 34 | 39
Completed | 34 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1-medication Pre and Post Procedure | Arm 2-Randomized to Placebo | Total
Number analyzed (Participants) | 34 | 39 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 39 | 73
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (17) | 46 (12) | 48 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 34 | 39 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Post-ERCP Pancreatitis Cases in Participants Who Are Administered Aprepitant and Placebo Prior to ERCP and One Day After ERCP:Assess the Total Number of Incidents of Post-ERCP Pancreatitis in Each Group (Treatment and Control).
Time Frame: 48 hours
Population: The number of participants who received the aprepitant or placebo were evaluated for ERCP pancreatitis. Each case of ERCP pancreatitis was tracked for the participant.
Measure: Number; unit: cases of ERCP in participants
Arm/Group | Arm 1-medication Pre and Post Procedure | Arm 2-Randomized to Placebo
Number analyzed (Participants) | 34 | 39
cases of ERCP in participants | 7 [1 to 73] | 7 [1 to 73]

2. Secondary Outcome: Incidence of Pain Post-ERCP, Within 48 Hours of ERCP, and at 1 Week Post-ERCP; Unrelated to Pancreatitis
Time Frame: 48 hours post ERCP and 1 week post ERCP
Population: There are 2 telephone assessments that participants are required to complete in order to analyze the outcome measure. The study team was unable to collect both assessments within the required timeframe due missed calls & lack of return calls from participants. Therefore data collection and analysis could not be completed per protocol.
Arm/Group | Arm 1-medication Pre and Post Procedure | Arm 2-Randomized to Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Who Were Hospitalized Within 7 Days Post-ERCP for Abdominal Pain That Did Not Meet Criteria for Acute Pancreatitis
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Arm 1-medication Pre and Post Procedure | Arm 2-Randomized to Placebo
Number analyzed (Participants) | 34 | 39
participants | 6 | 9

ADVERSE EVENTS:
Arm/Group | Arm 1-medication Pre and Post Procedure | Arm 2-Randomized to Placebo
Serious Adverse Events (participants affected / at risk) | 7/34 | 7/39
Other Adverse Events (participants affected / at risk) | 0/34 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-medication Pre and Post Procedure (N=34) | Arm 2-Randomized to Placebo (N=39)
ERCP pancreatitis (Endocrine disorders) | 7 (7) | 7 (7)

LIMITATIONS AND CAVEATS:
Unable to control for pre-procedure dosing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No